CLINICAL TRIAL: NCT06186284
Title: Impact of Technical Aids in the Occurrence of Carpal Tunnel Syndrome in Patients Undergoing Rehabilitation
Brief Title: Impact of Walking Aids on the Occurrence of Carpal Tunnel Syndrome in Rehabilitation
Acronym: CRUTCH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Valida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 23-001; 2023/17JAN/025 (Other: Comité d'éthique hospitalo-facultaire Saint-Luc -UCLouvain)
Record Dates: First submitted 2023-12-15; First posted 2023-12-29 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Carpal Tunnel Syndrome
Keywords: carpal tunnel
MeSH Terms: conditions — Carpal Tunnel Syndrome; Median Neuropathy | interventions — Nerve Conduction Studies

STUDY DESIGN:
Intervention Model Description: cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patient (Other): Rehabilitation patients using a technical walking aid will be followed up for development of carpal tunnel syndrome
  Interventions: Diagnostic Test: nerve conduction study; Diagnostic Test: ultrasonography wrists; Diagnostic Test: Boston carpal tunnel questionnaire; Diagnostic Test: clinical provocative tests for carpal tunnel syndrome

INTERVENTIONS:
Diagnostic Test: nerve conduction study — sensory and motor nerve conduction study of both median nerves and ulnar nerves
Diagnostic Test: ultrasonography wrists — assess the cross-sectional area of the median nerves and the ulnar nerves
Diagnostic Test: Boston carpal tunnel questionnaire — assess the severity of symptoms and the functional impact related to carpal tunnel syndrome
Diagnostic Test: clinical provocative tests for carpal tunnel syndrome — Tinel and Phalen's test to evaluate the presence of carpal tunnel syndrome

SUMMARY:
The purpose of this study is to assess the impact of the use of technical walking aids in the adult population undergoing rehabilitation by evaluating clinical, electrophysiological, and iconographic parameters before and after the use of these devices.

DETAILED DESCRIPTION:
The current evidence indicates that the short-term use of walking aids elicits pressure-induced anatomical changes of the median nerve and that long-term use of walking aids leads to a significant percentage of stroke patients developing clinical symptoms of carpal tunnel syndrome. We will investigate the consequences of using technical walking aids for gait in a broader population of rehabilitation patients. The rehabilitation setting per se may be considered a useful clinical 'human pathological model' for peripheral nerve entrapment. Recruited patients will be naïve to previous use of walking aids and de novo will start using them for gait rehabilitation, regardless of the underlying disease. This intervention model will allow us to identify clinical, electrophysiological, and anatomical changes of the median nerve due to the daily direct pressure elicited by walking aids. We consider that a one-month duration of use of walking aids is needed to observe detectable changes in electrophysiological and ultrasonographical assessment to elicit entrapment neuropathies in patients prone to developing them.

ELIGIBILITY:
Inclusion Criteria:

* admitted into an in-patient rehabilitation unit
* Functional Ambulation Category ≥ 1
* de novo need for a walking aid
* at least one functional upper limb
* expected duration of need for walking aid at least one month

Exclusion Criteria:

* less than 18 years old
* current use of walking aid or use of a walking aid less than 6 months ago)
* difficulty filling out questionnaires or understanding instructions in French
* medical contraindications to the use of walking aids
* refusal to sign the consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Boston Carpal Tunnel Questionnaire | one month
  The Boston Carpal Tunnel Questionnaire comprises two separate scales: the Symptom Severity Scale (SSS), which consists of 11 questions, and the Functional Status Scale (FSS), which consists of 8 items and requires respondents to score the difficulty of each item on a five-point scale. A final score is calculated for each scale (the sum of the individual scores divided by the number of items) and ranges from 1 to 5, with a higher score indicating a more severe handicap.

SECONDARY OUTCOMES:
PADUA score | one month
  The PADUA score is a classification of the neurophysiological severity of median neuropathy across the wrist. It is scored in 6 classes (1 to 6) with a higher score indicating greater neurophysiological damage to the median nerve
cross-sectional area of median nerve on ultrasound | one month
  Describes the diameter of the median nerve
clinical provocative tests of the median nerve | one month
  Tinel and Phalen's sign
Need for treatment of carpal tunnel syndrome | one month
  number of injections in the carpal tunnel/splinting of the wrist
cross-sectional area of ulnar nerve on ultrasound | one month
  describes the diameter of the ulnar nerve
amplitude of sensory nerve potential of the ulnar nerve | one month
  describes the functional status of the sensory ulnar nerve

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Parein, MD, Principal Investigator — Centre Hospitalier Valida; Patricia Dessart, MD, Study Director — Centre Hospitalier Valida; Samar M Hatem, MD,¨PhD, Study Chair — Centre Hospitalier Valida
Locations (1):
- Centre Hospitalier Valida, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No